CLINICAL TRIAL: NCT01696175
Title: Lactate Levels and Venous Oxygen Saturation in Children Admitted to a Dutch PICU
Brief Title: PICU Admission Lactate and Central Venous Oxymetry Study
Acronym: PALVOS
Status: Terminated | Type: Observational
Why Stopped: Researcher stopped activity at institution
Sponsor: Radboud University Medical Center (Other)
Collaborators: The Dutch Network of Excellence for Pediatric Intensive Care Research (Unknown)
Responsible Party: Principal Investigator, Joris Lemson, Medical director pediatric intensive care unit, Radboud University Medical Center
Other Study IDs: PALVOS
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Shock
Keywords: ScvO2; venous; oxymetry; lactate; children; PICU; Admission parameters of shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PICU admittance: Children equipped with an arterial and a central venous catheter within 12 hours after admittance to a Dutch PICU

SUMMARY:
Observational multicentre cohort study. Children admitted to a Dutch PICU are studied for lactate levels and ScvO2. Children instrumented with arterial and central venous catheters are included within the first 12 hours after admittance.

DETAILED DESCRIPTION:
Rationale: Hemodynamic therapy in children with circulatory insufficiency requires the use of hemodynamic monitoring parameters including parameters that reflect tissue/organ oxygenation and oxygen utilization. Two parameters are readily available at the bedside that may reflect this: arterial lactate level and central venous oxygen saturation (ScvO2). To date is it unknown if these parameters are useful in guiding treatment of critically ill children. Also it is unknown how often lactate and ScvO2 are abnormal in children admitted to a Dutch PICU or if they are related to each.

Objective: The objective of this study is to find the incidence of a raised lactate level and or a decreased ScvO2, to study their mutual relation and to study the relation between lactate, ScvO2 and outcome parameters in children admitted to a Dutch PICU.

Study design: Observational cohort study

Study population: children admitted to a PICU <= 16 years

Intervention (if applicable): No intervention

Main study parameters/endpoints: Arterial lactate level, central venous oxygen saturation (ScvO2), arterial blood gas analysis and general hemodynamic variables in the first 24 hours after admission. Parameters for organ dysfunction, severity of illness and outcome parameters like length of PICU stay.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: This is a strict observational design. No blood samples are taken for the purpose of this study. No intravascular catheters are inserted for the purpose of this study. No treatment strategy is associated with this study.

ELIGIBILITY:
Inclusion Criteria:

* Al children admitted to a PICU <= 16 years equipped with an arterial and central venous catheter in situ at admission or inserted within < 12 hours after admission to the PICU

Exclusion Criteria:

* Patients without an arterial or central venous catheter > 12 hours after of admission
* Patients with a known underlying metabolic disorder causing an elevated lactate level
* Patients with asthma and therapy (nebulized or intravenous) with salbutamol.
* Patients with an intoxication causing elevated lactate levels
* Premature children (<38 weeks GA)
* Patients on ECMO

Ages: 1 Week to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Al children admitted to a PICU <= 16 years equipped with an arterial and central venous catheter in situ at admission or inserted within < 12 hours after admission to the PICU.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-09; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
What is the incidence of a decreased ScvO2 and or a raised lactate level in children admitted to Dutch PICU's in the first 24 hours after admission to the PICU | first 24 hours after admission
  What is the incidence of a decreased ScvO2 and or a raised lactate level in children admitted to Dutch PICU's in the first 24 hours after admission to the PICU

CONTACTS AND LOCATIONS:
Locations (1):
- RUNMC, Nijmegen, Netherlands